CLINICAL TRIAL: NCT06177743
Title: Evaluation of Effectiveness and Safety of Coroflex ISAR NEO Stent in Routine Clinical Practice; A Multicenter, Prospective Observational Study
Brief Title: IRIS-Coroflex NEO Cohort
Acronym: IRIS Coroflex
Status: Recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: The CardioVascular Research Foundation (CVRF) (Unknown)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2023-05
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Stenosis; Coronary Artery Disease
Keywords: percutaneous coronary intervention
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coroflex ISAR NEO: Patients receiving percutaneous coronary intervention with Coroflex ISAR NEO stents
  Interventions: Device: Coroflex ISAR NEO stent

INTERVENTIONS:
Device: Coroflex ISAR NEO stent — Percutaneous coronary intervention with Coroflex ISAR NEO stent

SUMMARY:
The objective of this study is to evaluate the effectiveness and safety of Coroflex ISAR NEO stents in comparison to other drug-eluting stents (DES) in real-world practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 19 years old
2. Patients receiving Coroflex ISAR NEO stents.
3. The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.

Exclusion Criteria:

1. Patients with a mixture of other DESs
2. Terminal illness with life expectancy <1 year.
3. Patients with cardiogenic shock

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving Coroflex ISAR NEO stents.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
the composite of death, nonfatal myocardial infarction (MI), or ischemic-driven Target- Vessel Revascularization (TVR) | 12 months
  the composite of death, nonfatal myocardial infarction (MI), or ischemic-driven Target- Vessel Revascularization (TVR) at 12 months post procedure.
  A composite endpoint is an endpoint that is a combination of multiple clinical endpoints. An event is considered to have occurred if any one of several different events is observed.

SECONDARY OUTCOMES:
the event rate of all cause death | 5 years
the event rate of cardiac death | 5 years
the event rate of myocardial infarction | 5 years
the composite event rate of death, or myocardial infarction (MI) | 5 years
the composite event rate of cardiac death, or myocardial infarction (MI) | 5 years
the event rate of Target- Vessel Revascularization (TVR) | 5 years
the event rate of Target- lesion Revascularization (TLR) | 5 years
the event rate of stent thrombosis | 5 years
  according to an Academic Research Consortium (ARC) criteria
the event rate of stroke | 5 years
the event rate of Procedural success | 5 days
  defined as achievement of a final diameter stenosis of <30% by visual estimation, without the occurrence of death, Q-wave MI, or urgent revascularization during the index hospitalization.

CONTACTS AND LOCATIONS:
Locations (11):
- South Korea (11):
  - Asan Medical Center, Seoul, Songpa-gu
  - Bucheon Sejong Hospital, Bucheon-si
  - The Catholic Univ. of Korea BUCHEON ST.Mary's hospital, Bucheon-si
  - Veterans Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Inje University Ilsan Paik Hospital, Ilsan
  - Myongji Hospital, Ilsan
  - Sejong Chungnam National University Hospital, Sejong
  - Seoul National University Boramae Medical Center, Seoul
  - The Catholic university of Korea, ST. Vincent's Hospital, Suwon
  - Uijeongbu Eulji Medical Center, Uijeongbu-si

IPD SHARING:
Plan to Share IPD: Undecided